CLINICAL TRIAL: NCT02172664
Title: Clinical Evaluation of a Universal Adhesive in Noncarious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Jeffrey A. Platt, Associate Professor of Dental Materials, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVOC2014
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Cervical Lesions
Keywords: noncarious cervical lesions; dental adhesive; retention; enamel margin discoloration; self etch; selective etch procedures
MeSH Terms: interventions — Ivoclar Universal Cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhese Universal with self etch enamel etching (Active Comparator): patients will receive one restoration on randomly selected study tooth utilizing the self-etch universal adhesive (Adhese Universal, Ivoclar Vivadent) with no separate enamel etching
  Interventions: Procedure: Self etch enamel etching; Procedure: selective etch protocol; Device: Adhese Universal
- selective etch protocol followed by Adhese Universal (Experimental): patients will receive one restoration on randomly selected study tooth utilizing a 37% phosphoric acid solution followed by application of self-etch universal adhesive (Adhese Universal, Ivoclar Vivadent)
  Interventions: Procedure: Self etch enamel etching; Procedure: selective etch protocol; Device: Adhese Universal

INTERVENTIONS:
Procedure: Self etch enamel etching — The adhesive will be applied according to manufacturer's instructions. If the lesion is greater than 2 mm in any dimension, incremental placement of Tetric EvoCeram composite (Ivoclar Vivadent) will occur with the first increment being placed against enamel.
  Other Names: Adhese Universal; Ivoclar Vivadent
Procedure: selective etch protocol — Total Etch (37% phosphoric acid; Ivoclar) will be placed on the enamel margin with no intentional placement on the dentin within the lesion. The adhesive will then be applied as instructed by the manufacturer. Tetric EvoCeram composite will be placed, light-cured, finished, and polished in the same manner as for the self-etch group.
Device: Adhese Universal — the universal adhesive, Adhese Universal , will be applied to the selected tooth following manufacturer instructions

SUMMARY:
The purpose of this prospective clinical trial will be to evaluate the efficacy of an FDA approved and marketed universal dental adhesive formulation in adult noncarious cervical lesions using self-etch and selective etch approaches.

The hypothesis is that using a selective enamel etch with this universal adhesive will enhance the restoration margin performance.

DETAILED DESCRIPTION:
The purpose of this prospective clinical trial will be to evaluate the efficacy of a newly formulated universal dental adhesive formulation in adult noncarious cervical lesions using self-etch and selective etch approaches.

Thirty-three patients with at least two non-carious cervical lesions will receive one restoration utilizing the self-etch universal adhesive with no separate enamel etching and another restoration utilizing the universal adhesive and a a selective etch protocol in which in which enamel is etched with 37% phosphoric acid.

After a screening/baseline visit at which the restorative procedures listed above will conducted, the patient will be seen at recall visits after approximately 6, 12 and 24 months to observe sensitivity, retention, marginal discoloration and marginal adaptation.

ELIGIBILITY:
Inclusion Criteria:

* 1.1. Inclusion criteria

  1. Willing to provide written consent and authorization for participation.
  2. Be between 20 and 75 years of age at the time of recruitment
  3. Have at least two non-carious cervical lesions present in canine or premolar teeth;
  4. Anticipates availability for recalls (roughly 6 month, 12 month, and 24 month) through the two-year study period
  5. The lesions selected will be at least 1 mm in depth (measured with a perio probe) and contain both enamel and dentin margins.

     Exclusion Criteria:

1.2. Exclusion criteria

1. Severe medical complications (organ transplants, cancer, immunocompromised, long term antibiotic or steroid therapy);
2. Active caries on study teeth;
3. Bleeding on probing of study teeth;
4. Generalized severe periodontitis;
5. Patient reported symptoms (burning mouth, loss or diminished taste, saliva amount too little, needs liquids to eat dry foods) or clinical signs (erythematous tongue, chelitis, lack of pooled saliva) associated with dry mouth;
6. Patients determined to be at a high risk of caries as determined by a Caries Risk Assessment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Platt, DDS, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Non-carious cervical lesions
Period: Overall Study
Arm/Group | Adhese Universal With Self Etch Enamel Etching | Selective Etch Protocol Followed by Adhese Universal
Started | 33; 40 Non-carious cervical lesions | 33; 41 Non-carious cervical lesions
Completed | 27; 35 Non-carious cervical lesions | 27; 31 Non-carious cervical lesions
Not Completed | 6; 5 Non-carious cervical lesions | 6; 10 Non-carious cervical lesions
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 1 | 1
Not completed — Moved out of area | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received both interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Customized [Count of Participants; unit: Participants]
  20-39 | 4
  40-59 | 14
  60+ | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Retention of Restorations
Description: The primary outcome measure will be restoration retention. In these non-retentive dental lesions, the adhesive will be the only mode of retention. Failure of the adhesive would result in loss of the restoration.
Time Frame: 6, 12, 24 months
Population: Available number of participants at each time point are reported.
Measure: Count of Units; unit: Non-carious cervical lesions
Units Other Than Participants: Non-carious cervical lesions
Arm/Group | Adhese Universal With Self Etch Enamel Etching | Selective Etch Protocol Followed by Adhese Universal
Number analyzed (Participants) | 33 | 33
Number analyzed (Non-carious cervical lesions) | 40 | 41
Non-carious cervical lesions
  6 months: number analyzed (Participants) | 31 | 31
  6 months: number analyzed (Non-carious cervical lesions) | 38 | 38
  6 months | 38 | 38
  12 months: number analyzed (Participants) | 30 | 30
  12 months: number analyzed (Non-carious cervical lesions) | 37 | 37
  12 months | 37 | 37
  24 months: number analyzed (Participants) | 27 | 27
  24 months: number analyzed (Non-carious cervical lesions) | 35 | 31
  24 months | 34 | 31

2. Secondary Outcome: Number of Restoration Margins Marked as Stained or Discolored
Description: The secondary outcome measure was the presence of discoloration of restoration margins as determined by blinded evaluators.
Time Frame: 6, 12, 24 months
Population: Available number of participants at each time point are reported.
Measure: Count of Units; unit: Non-carious cervical lesions
Units Other Than Participants: Non-carious cervical lesions
Arm/Group | Adhese Universal With Self Etch Enamel Etching | Selective Etch Protocol Followed by Adhese Universal
Number analyzed (Participants) | 33 | 33
Number analyzed (Non-carious cervical lesions) | 40 | 41
Non-carious cervical lesions
  6 months: number analyzed (Participants) | 31 | 31
  6 months: number analyzed (Non-carious cervical lesions) | 38 | 38
  6 months | 1 | 1
  12 months: number analyzed (Participants) | 30 | 30
  12 months: number analyzed (Non-carious cervical lesions) | 37 | 37
  12 months | 0 | 0
  24 months: number analyzed (Participants) | 27 | 27
  24 months: number analyzed (Non-carious cervical lesions) | 35 | 31
  24 months | 5 | 1

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were not monitored per intervention.
Groups:
- All Study Participants: Adverse events were not monitored per intervention.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02172664/Prot_SAP_000.pdf